CLINICAL TRIAL: NCT06764823
Title: Evaluation of the Effect of Intracanal Cryotherapy on Postoperative Pain After Retreatment: a Randomized Controlled Clinical Trial
Brief Title: Effect of Intracanal Cryotherapy on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Arzu Kaya Mumcu, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUTAHYAHSU-2
Record Dates: First submitted 2024-12-25; First posted 2025-01-08 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Retreatment; Cryotherapy
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: Experimental Group: The final irrigation solution will be 5 mL of 0.9% physiological saline solution at 2.5°C, irrigated for 5 minutes.
  Control Group: The final irrigation for the control group will be 5 mL of 0.9% physiological saline solution at room temperature, irrigated for 5 minutes.
Who Masked: Participant
Masking Description: The participants were not informed about the temperature of the saline solution applied to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryotherapy (Experimental): The final irrigation solution will be 5 mL of 0.9% physiological saline solution at 2.5°C, irrigated for 5 minutes.
  Interventions: Other: Cryotherapy
- Control (Other): The final irrigation for the control group will be 5 mL of 0.9% physiological saline solution at room temperature, irrigated for 5 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Other: Cryotherapy — In the cryotherapy group, after completing the biomechanical preparation, the root canals will be irrigated with 5 mL of 0.9% physiological saline solution at 2.5°C for 5 minutes; the solution will be stored in the refrigerator until use.
  Arms: Cryotherapy
Other: Control — In the control group, the final irrigation will be performed using 5 mL of 0.9% physiological saline solution at room temperature for 5 minutes.
  Arms: Control

SUMMARY:
Introduction: Since 1960, cryotherapy, involving the application of cold, has been used in various fields of medicine for pain treatment. Cold application induces three main physiological tissue responses: a decrease in metabolic activity, a reduction in blood flow, and the inhibition of neural receptors in the skin and subcutaneous tissues. Consequently, cryotherapy slows down neural signals and reduces the release of chemical mediators responsible for pain. Recently, the use of cryotherapy in root canal treatment, in the form of cold saline irrigation, has been investigated in several randomized controlled trials. The aim of this study is to evaluate the effect of cold saline irrigation as a final irrigant on postoperative pain following the biomechanical preparation of root canals in patients undergoing non-surgical retreatment.

Method: Sixty single-rooted, single-canal teeth requiring non-surgical root canal retreatment were randomly assigned to two groups (n = 30): a cryotherapy group and a control group. All the treatments were completed during a single visit. Protaper Universal Retreatment files (D1, D2, and D3) were used for the removal of gutta-percha and root canal preparation, and irrigation was performed using 2.5 % NaOCl and 17% EDTA. The cryotherapy group had a final irrigation temperature of 2.5 °C for 5 min before root canal obturation, whereas the control group received irrigation at room temperature.

All patients will be asked to record their postoperative pain levels on VAS scales at 6, 12, and 24 hours, and at 2, 3, and 7 days after treatment. Patients will be asked to rate the pain they experience during the 7-day postoperative period on a scale from 0 to 10. Statistical analysis was performed using the Chi-Square test, Mann-Whitney test, and Independent Samples test, with the significance level set at 0.05.

DETAILED DESCRIPTION:
Study design

To address the aim of the research, a prospective randomized clinical trial was designed. This study will be conducted at the Department of Endodontics, Oral and Dental Health Practice and Research Center, Faculty of Dentistry, Kütahya Health Sciences University.

Patients will be informed about the study design, and all participants will be asked to read and sign the informed consent form if they agree to participate. Patient forms including demographic information, medical history, and PAI scores will be filled out. Patients who meet the inclusion criteria and agree to participate will be randomly divided into two groups: the first group will receive routine retreatment and root canal therapy followed by intracanal cryotherapy, while the second group will receive routine retreatment and root canal therapy followed by room temperature saline solution.

Root Canal Treatment Procedure The sample size for the study was calculated using the G*Power statistical program (ver.3.1.9.7). Accordingly, with a power (test strength) of 0.85, an effect size of 0.8, and a type-1 error (α) of 0.05, the minimum number of patients/samples required for each group was determined to be 30, making a total of 60 patients. Patients will undergo a single visit retreatment. Root canal treatments will be performed by a single clinician following a standard protocol. After selecting an appropriate anesthesia technique for the tooth to be treated, 1.8 mL of 4% articaine with 1:200,000 epinephrine will be injected, followed by rubber dam isolation. After opening the access cavity, the existing root canal filling will be removed using Protaper Universal Retreatment files (D1, D2, and D3) and a VDW Gold endomotor according to the manufacturer's instructions, and the working length will be established with a size 15 K-file. The working length will be confirmed with periapical radiographs. No chemical solvents will be used in the removal of the root canal filling. A size 30 H-file will be used to clean the remnants of the root canal filling. The root canal preparation will then be completed using the WaveOne Gold file system size 45.05. Between files, the canals will be irrigated with 2.5% NaOCl using a 31 gauge side-vented needle, 2 mm short of the working length.

After completing the root canal preparation, final irrigation will be performed using passive ultrasonic irrigation activation with 5 mL of 2.5% NaOCl for 1 minute, followed by 5 mL of saline and then 2 mL of 17% EDTA for 1 minute. In the cryotherapy group, after completing the biomechanical preparation, the root canals will be irrigated with 5 mL of 0.9% saline solution at 2.5°C for 5 minutes; the solution will be kept in the refrigerator until use. In the control group, the final irrigation will be performed using 5 mL of 0.9% saline solution at room temperature for 5 minutes.

The root canals will then be dried with paper points, filled with root canal sealer, and obturated using the single cone technique appropriate for the final preparation size. The access cavity will be sealed with a temporary filling, and the patient will be scheduled for a follow-up appointment in 1 week. Patients will be reminded by phone to record their pain levels at specified hours and days, and to record any analgesic consumption (including dose and time). Patients who report taking analgesics will be excluded from the study. Patients will be asked to record their postoperative pain levels on VAS scales at 6, 12, and 24 hours, and at 2, 3, and 7 days after treatment. The results will be statistically analyzed. Statistical analysis was performed using the Chi-Square test, Mann-Whitney test, and Independent Samples test, with the significance level set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* No analgesic anti-inflammatory medication intake in the last 72 hours
* Age 18-59
* PAI score of 4 (well-defined periapical radiolucency)
* Previous root canal treatment 2-4 mm short
* At least 4 years since the existing root canal treatment
* Asymptomatic acute apical periodontitis requiring retreatment of single-rooted teeth

Exclusion Criteria:

* Medically compromised patients
* Pregnant patients
* Patients taking analgesic or anti-inflammatory medication
* Patients who refuse to participate
* Patients with an allergy to articaine
* Teeth with internal and external resorption
* Teeth with open apices

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Radiographic assessment of retreatment success | "0 hours" (Treatment appointment)
  The quality of endodontic treatment will be evaluated according to the criteria established by Cleen et al.: (a) Adequate: Root canal filling 0-2 mm short of the radiographic apex. (b) Inadequate: Root canal filling more than 2 mm short of the radiographic apex. (c) Inadequate: Root canal filling extending beyond the radiographic apex.
  The density of the root canal treatment will be assessed based on the criteria of Dugas et al.: (a) Adequate: Uniform radiopacity and tight adaptation of gutta-percha to the root canal walls. (b) Inadequate: Visible voids in the root canal or unfilled canals.
  For the retreatment to be considered successful, it must be rated as adequate according to both of the above criteria.

SECONDARY OUTCOMES:
Post-operative pain | 6., 12., 24. hours and 2., 3. and 7. day
  Secondary endpoint is the evaluation of the effect of intracanal cryotherapy on patients' postoperative pain, assessed using the visual VAS scale included in the treatment protocol.
  All patients will be asked to record their postoperative pain levels on VAS scales at 6, 12, and 24 hours, and at 2, 3, and 7 days after treatment. Patients will be asked to rate the pain they experience during the 7-day postoperative period on a scale from 0 to 10, where 0 represents no pain and 10 represents severe pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kutahya Health Sciences University Faculty of Dentistry, Kütahya
  - Kutahya Health Sciences University, Kütahya

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR